CLINICAL TRIAL: NCT03708809
Title: Immediate Versus Delayed Initiation of the 13.5 mg Levonorgestrel-releasing Intrauterine System Following Surgical Termination of Pregnancy
Brief Title: Immediate Versus Delayed Initiation of Intrauterine System
Acronym: JANESS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: could not be funded
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4671-17-SMC
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Contraception
Keywords: IUD, contraception, levonogestral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Immediate insertion (Experimental): The intrauterine system will be inserted immediately after surgical termination of pregnancy, before awakening from anesthesia
  Interventions: Device: Intrauterine system
- Delayed insertion (Experimental): The intrauterine system will be inserted on the first menstruation after termination of pregnancy. Women allocated to this arm will be asked to contact the study coordinator in order to visit the hospital on the proper timing for IUD insertion.
  Interventions: Device: Intrauterine system
- Control (Other): Women who refuse to actively participate in the intervention groups will be offered consultation on other options for contraception during gynecological clinic visit after fist menstruation from termination of pregnancy.
  Interventions: Other: Alternative contraception to intrauterine system

INTERVENTIONS:
Device: Intrauterine system — 13.5 mg levonorgestrel-releasing intrauterine system
  Other Names: Janess
  Arms: Delayed insertion; Immediate insertion
Other: Alternative contraception to intrauterine system — Alternative contraception including contraception pills, hormonal patches, hormonal vaginal , condomsring,
  Arms: Control

SUMMARY:
Contraception for teenagers and young adults presents a huge challenge for the clinician as more than half of all unintended pregnancies occur as a result of inconsistent or discontinued use of contraceptives . Possible solution is promoting the use of long acting reversible contraception, (LARC) among them the intrauterine device (IUD). IUD provide safe, highly effective, long-term contraception. Immediate IUD insertion after the termination of pregnancy (TOP) is a very convenient way to provide contraception as it is an opportune moment to carry out this short, easy, and safe procedure.

Janess is a T-shaped intrauterine delivery system that was introduced lately, which slowly releases a small amount (13.5 mg) of levonorgestrel after its installation inside the womb and provides contraception for up to three years.

The aim of this study to compare insertion of 13.5 mg levonorgestrel-releasing intrauterine system after surgical abortion immediately versus delayed insertion (at menstruation)

DETAILED DESCRIPTION:
The rate of repeat induced abortion varies from 30% to 38% in northern Europe. Young women, parous women and those with a history of abortion were found to be the main risk factors associated with recurrent termination of pregnancy. Young women may lack knowledge or access to conventional methods of preventing pregnancy, as they may be too embarrassed or frightened to seek such information. Contraception for teenagers and young adults presents a huge challenge for the clinician as more than half of all unintended pregnancies occur as a result of inconsistent or discontinued use of contraceptives . Possible solution is promoting the use of long acting reversible contraception, (LARC) among them the intrauterine device (IUD), that was found well suited even for adolescents. Because IUDs do not require active use once they have been inserted, and have a very low failure rate, their increased use has the potential to substantially reduce unintended pregnancies. IUD provide safe, highly effective, long-term contraception, but they are underused.

Immediate initiation of any contraceptive method after an abortion has been linked to a reduced risk of repeat abortion. Immediate IUD insertion after the termination of pregnancy (TOP) is a very convenient way to provide contraception as it is an opportune moment to carry out this short, easy, and safe procedure. As the cervix is dilated, insertion is virtually painless. Following insertion, the woman is protected immediately, before ovulation returns, usually within 7-10 days after first-trimester abortion.

Lately, a new intrauterine device directed for young women was introduced. It is a T-shaped intrauterine delivery system which slowly releases a small amount (13.5 mg) of levonorgestrel after its installation inside the womb. The system is intended for contraception for a period of up to 3 years. It works by reducing the monthly growth of the lining of the womb and thickening of the cervical mucosal layer.

To the best of the investigator's knowledge this is the first study to compare insertion of 13.5 mg levonorgestrel-releasing intrauterine system after surgical abortion immediately versus delayed insertion (at menstruation) .

ELIGIBILITY:
Inclusion Criteria:

* Women that are about to go through surgical termination of first trimester pregnancy
* Age ≥ 18 years
* Nulliparous

Exclusion Criteria:

* structural uterine abnormality
* submucosal fibroids
* suspected uterine or cervical neoplasia
* acute pelvic inflammatory disease
* acute liver disease or previous breast cancer

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Continuation rate after one year from insertion | estimated time of one year follow up from insertion

SECONDARY OUTCOMES:
Expulsion rate | On first visit after menstruation from insertion, 3 month from insertion and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr Sasson, M.D, Principal Investigator — Sheba Medical Center, Tel-Hashomer
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heikinheimo O, Gissler M, Suhonen S. Age, parity, history of abortion and contraceptive choices affect the risk of repeat abortion. Contraception. 2008 Aug;78(2):149-54. doi: 10.1016/j.contraception.2008.03.013. Epub 2008 May 27. PMID 18672117
- [Result] Apter D. Contraception options: Aspects unique to adolescent and young adult. Best Pract Res Clin Obstet Gynaecol. 2018 Apr;48:115-127. doi: 10.1016/j.bpobgyn.2017.09.010. Epub 2017 Sep 28. PMID 29032945
- [Result] Hubacher D, Cheng D. Intrauterine devices and reproductive health: American women in feast and famine. Contraception. 2004 Jun;69(6):437-46. doi: 10.1016/j.contraception.2004.01.009. PMID 15157788
- [Result] Goodman S, Hendlish SK, Reeves MF, Foster-Rosales A. Impact of immediate postabortal insertion of intrauterine contraception on repeat abortion. Contraception. 2008 Aug;78(2):143-8. doi: 10.1016/j.contraception.2008.03.003. Epub 2008 May 14. PMID 18672116
- [Result] Lahteenmaki P, Luukkainen T. Return of ovarian function after abortion. Clin Endocrinol (Oxf). 1978 Feb;8(2):123-32. doi: 10.1111/j.1365-2265.1978.tb02160.x. PMID 630723